CLINICAL TRIAL: NCT01661868
Title: Phase II Study of Single Agent Olaparib for Patients With Recurrent BRCA Deficient Ovarian Cancer With No Prior PARP Exposure or Prior PARP Inhibitor Exposure
Brief Title: Olaparib for Patients With Recurrent BRCA Deficient Ovarian Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Drug not available.
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Ursula A. Matulonis, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11-170
Record Dates: First submitted 2011-10-24; First posted 2012-08-10 (Estimated); Last update posted 2012-08-21 (Estimated); Status verified 2012-08

CONDITIONS: Ovarian Cancer; Peritoneal Cancer; Fallopian Tube Cancer
Keywords: BRCA1 mutation; BRCA2 mutation
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms | interventions — olaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PARP Inhibitor Naive (Active Comparator): Patients with no prior PARP inhibitor treatment
  Interventions: Drug: Olaparib
- Prior PARP Inhibitor (Active Comparator): Patients previously treated with a PARP inhibitor other than olaparib
  Interventions: Drug: Olaparib

INTERVENTIONS:
Drug: Olaparib — Tablet formulation will be used.
  Other Names: AZD2281

SUMMARY:
This research study is a way of gaining new knowledge about a drug called olaparib in women who have either: 1)never received a PARP inhibitor before to treat ovarian cancer (group 1) or 2)participants who have received a PARP inhibitor before to treat ovarian cancer, with the exception of olaparib (group 2). PARP inhibitors are drugs tht prevent cancer cells from repairing their DNA. In this research study, we are looking to see how well the drug olaparib works in women who have never received a PARP inhibitor for recurrent ovarian cancer as well as those who have received a prior PARP inhibitor and whose cancer has re-grown after receiving that PARP inhibitor.

DETAILED DESCRIPTION:
Olaparib tablets will be taken twice daily, orally, in treatment cycles lasting 4 weeks.

On days 1, 8, 12 and 22 of the first 2 cycles and day 1 of all other cycles, subjects will have a physical exam, be asked questions about their general health, and specific questions about any problems they might be having and any medications they are taking.

Tumor will be assess by either CT or MRI scan every 2 cycles (every 2 months). Tumor biopsies will be optional in this study. Only participants that have received a PARP inhibitor in the past will be asked to have a biopsy of their tumor.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed ovarian, peritoneal or fallopian tube cancer that has recurred following a platinum-based regimen used at initial diagnosis
* Measurable disease
* Estimated life expectancy greater than 16 weeks
* Normal organ and marrow function
* Evidence of non-childbearing status for women of childbearing potential
* Able to swallow oral medication

Exclusion Criteria:

* Pregnant or breastfeeding
* Prior PARP inhibitor use for another cancer such as breast cancer
* Receiving any other study agents or any other anti-cancer treatment
* Known brain metastases
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to olaparib
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive hear failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* History of a different malignancy unless disease-free for at least 5 years
* Currently experiencing seizures or currently being treated with any anti-epileptic for seizures
* Human immunodeficiency virus (HIV) positive on combination antiretroviral therapy
* Presence of gastrointestinal disorders that, in the investigator's opinion, are likely to interfere with the absorption of olaparib, or with the patient's ability to take regular oral medication

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-08; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Response Rates | 1 year
  To determine the RECIST 1.1. response rates of the oral PARP inhibitor olaparib based on prior exposure of a PARP inhibitor; patients who have received and subsequently have had disease progression with a prior PARP inhibitor versus no prior exposure to a PARP inhibitor in patients with germline BRCA mutations who have recurrent ovarian, fallopian tube or peritoneal cancer who have measurable cancer.

SECONDARY OUTCOMES:
Toxicity | 1 year
  Assess toxicity profile of olaparib according to the Common Terminology Criteria for Adverse Events (CTCAE, version 4)
Progression free survival | 1 year
  Assess progression free survival (PFS) and 6 month PFS rate
Response Rate | 1 year
  Assess CA125 response rate

CONTACTS AND LOCATIONS:
Overall Officials: Ursula A Matulonis, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States